CLINICAL TRIAL: NCT05573919
Title: VivAer: A Correlation Between Symptom Scores and Objective Findings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Auddie Sweis, Principal Investigator, Endeavor Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EH22-177
Record Dates: First submitted 2022-10-04; First posted 2022-10-10 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Nasal Obstruction; Medically Unexplained Symptoms; Airway Obstruction; Airway Remodeling
Keywords: VivAer; Symptom Improvement
MeSH Terms: conditions — Nasal Obstruction; Medically Unexplained Symptoms; Airway Obstruction; Airway Remodeling

STUDY DESIGN:
Intervention Model Description: Patients who are to undergo the VivAer procedure for nasal obstruction with Dr. Auddie Sweis or Dr. Joseph Raviv will be recruited to this study. They will be issued questionnaires and have PNIF measurements taken to assess their symptoms before and after the procedure in order to determine the objective improvement in the patients' symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- VivAer Patients (Experimental): These patients will undergo the VivAer procedure, which involves the use of a stylus to deliver radiofrequency heating to the nasal sidewall to reshape the tissue. This will be done to resolve the patients' nasal obstruction. They will have PNIF measurements taken and will complete symptom assessment questionnaires before and after the VivAer procedure.
  Interventions: Device: VivAer Stylus

INTERVENTIONS:
Device: VivAer Stylus — This device will be used to complete its corresponding procedure, which involves reshaping a patient's nasal sidewall tissue through the delivery of radiofrequency heating.

SUMMARY:
This is a prospective, single-center study. This study seeks to determine the objective improvement in nasal airflow in patients after undergoing the VivAer procedure, which involves the use of a stylus to deliver controlled and targeted low energy radiofrequency heating (heating by applying high-frequency radio waves) to the nasal sidewall to gently reshape the tissues. Patients who experience refractory, or medically unexplained, nasal obstruction often have symptoms that are not alleviated or resolved by standard non-surgical treatment options. VivAer, a recently developed, FDA-approved procedure, is one of the standard surgical treatments for nasal obstruction. Unlike most of the other established surgical treatments for nasal obstruction, however, VivAer is a minimally-invasive procedure, and it is an outpatient intervention that can be performed under local anesthetic. Eligible patients who are enrolled in the study will undergo the VivAer procedure, and will return to the clinic for three in-office follow-up visits at 4, 12, and 24 weeks after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older seeking treatment for nasal obstruction and willing to undergo an office-based procedure.
* Nasal obstruction, defined as ≥60 by the NOSE scale.
* The nasal valve is the primary or significant contributor to the subject's nasal obstruction as determined by the investigator, based on clinical presentation, physical examination, or nasal endoscopy.
* Subjects has symptomatic improvement with use of external or internal nasal dilators, Q-Tip or curette test (manual intranasal lateralization), or the Cottle Maneuver (manual lateral retraction of the cheek).
* Subject experienced minimal symptomatic improvement after the four-week fluticasone steroid nasal spray regimen.

Exclusion Criteria:

* Prior surgery to the nasal valve, rhinoplasty, septoplasty, inferior turbinate reduction or other surgical nasal procedures within the past 12 months.
* Severe and/or chronic sinusitis, recurrent sinusitis, or allergies leading to nasal obstruction and currently requiring oral corticosteroid therapy.
* Severe case of any of the following; septal deviation, turbinate hypertrophy, polyps, or ptotic nasal tip believed to be the primary contributor to the subject's nasal obstruction symptoms and warranting surgical intervention.
* Known or suspected allergies or contraindications to the anesthetic agents and/or antibiotic medications to be used during the study procedure session.
* Known or suspected pregnancy, or lactation.
* Other medical conditions that the investigator believed would predispose subject to poor wound healing or increased surgical risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
PNIF Measurement | This will be administered before the VivAer procedure and at 4, 12, and 24 weeks post procedure.
  The change in the severity of the patients' nasal obstruction will be measured using a Peak Nasal Inspiratory Flow (PNIF) meter. This meter measures nasal patency by measuring the volume of air that is inhaled per minute during normal breathing.

SECONDARY OUTCOMES:
NOSE Score | This will be administered before the VivAer procedure and at 4, 12, and 24 weeks post procedure.
  The patients will self-assess the degree of their symptoms with the Nasal Obstructive Symptom Evaluation (NOSE) questionnaire. The questionnaire consists of 5 questions ranking the severity of one's symptoms on a scale of 0-5. The responses are summed and multiplied by 20 to generate a symptom score out of 0-100. Higher scores indicate worse outcomes.
SNOT-22 Score | This will be administered before the VivAer procedure and at 4, 12, and 24 weeks post procedure.
  The patients will self-assess the degree of their symptoms with the SinoNasal Outcome Test (SNOT-22) questionnaire. The questionnaire consists of 22 questions ranking the impact of a patient's symptoms on their quality of life on a scale of 0-5. The responses are summed to generate a score out of 110. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Auddie Sweis, MD, Principal Investigator — Endeavor Health; Joseph Raviv, MD, Principal Investigator — Endeavor Health
Locations (2):
- United States (2):
  - Swedish Covenant Hospital, Chicago, Illinois
  - NorthShore Skokie Hospital, Skokie, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobowitz O, Driver M, Ephrat M. In-office treatment of nasal valve obstruction using a novel, bipolar radiofrequency device. Laryngoscope Investig Otolaryngol. 2019 Feb 4;4(2):211-217. doi: 10.1002/lio2.247. eCollection 2019 Apr. PMID 31024989
- [Background] Ephrat M, Jacobowitz O, Driver M. Quality-of-life impact after in-office treatment of nasal valve obstruction with a radiofrequency device: 2-year results from a multicenter, prospective clinical trial. Int Forum Allergy Rhinol. 2021 Apr;11(4):755-765. doi: 10.1002/alr.22667. Epub 2020 Aug 9. PMID 32810380
- [Background] Stewart MG, Smith TL, Weaver EM, Witsell DL, Yueh B, Hannley MT, Johnson JT. Outcomes after nasal septoplasty: results from the Nasal Obstruction Septoplasty Effectiveness (NOSE) study. Otolaryngol Head Neck Surg. 2004 Mar;130(3):283-90. doi: 10.1016/j.otohns.2003.12.004. PMID 15054368
- [Background] Lipan MJ, Most SP. Development of a severity classification system for subjective nasal obstruction. JAMA Facial Plast Surg. 2013 Sep-Oct;15(5):358-61. doi: 10.1001/jamafacial.2013.344. PMID 23846399

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT05573919/Prot_SAP_000.pdf